CLINICAL TRIAL: NCT00747240
Title: Platelet-activating Factor Acetylhydrolase (Paf-ah) Gene Expression And The Incidence Of Chronic Lung Disease (Cld) In Very Low Birth Weight Infants
Brief Title: Platelet-activating Factor Acetylhydrolase (Paf-ah) Gene Expression
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Christian Con Yost, University of Utah
Other Study IDs: 00008854
Record Dates: First submitted 2008-09-03; First posted 2008-09-05 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2014-07

CONDITIONS: Low Birth Weight Infant
Keywords: Ile198Thr; Ala379Val; variants; PAF-AH

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective observational study to determine whether there is an association between the presence of platelet-activating factor acetylhydrolase (PAF-AH) gene polymorphisms and the development of chronic lung disease in very low birth wight infants. Infants < 1500 grams at birth who require mechanical ventilation will be enrolled in the first 5 days of life after obtaining informed consent. A total of 1 ml of blood will be drawn and utilized for isolation of DNA for genotyping and for measurement of PAF-AH activity in serum.

DETAILED DESCRIPTION:
Chronic lung disease (CLD) is a frequent and severe complication of premature birth. Between 3,000 and 7,000 infants develop CLD per year in the United States [6, 7]. Mortality rates for infants with CLD vary from 5% to 30% [8, 9]. Despite recent advances in neonatal care the incidence of CLD has not decreased, likely due to the survival of smaller more immature infants. Current therapies for CLD, many with demonstrated short-term but not long-term efficacy, include diuretics, bronchodilators, and corticosteroids. No therapeutic study published to date has demonstrated any single medication or combination of medication that improves survival or dramatically decreases severity or duration of illness.

The specific mechanism(s) that lead to CLD have not been clearly defined, but it is likely that multiple factors contribute to the disease. The most important factors that have been implicated, directly or indirectly, are prematurity, barotrauma, oxygen toxicity, inflammation and infection [7 ]. Although barotrauma and oxygen toxicity may directly injure the immature lung, recruitment and activation of inflammatory cells may potentiate lung damage and impaired healing. Several studies have shown persistent elevation of neutrophils, alveolar macrophages and high concentrations of lipid mediators in the tracheal effluent from infants with CLD [7]. Activated inflammatory cells in the lung may release products that alter pulmonary function and / or damage lung tissue leading to pulmonary edema, airway hyper-reactivity, and pulmonary hypertension which are pathophysiologic characteristics of infants with chronic lung disease [10].

Activated neutrophils and macrophages secrete platelet-activating factor (PAF). PAF is a phospholipid with diverse, potent physiologic activities. Many of the pathophysiologic abnormalities of CLD correlate with the actions of PAF. For example, PAF increases vascular permeability, which could lead to pulmonary edema. PAF causes bronchoconstriction and vascular smooth muscle constriction that could lead to the increased airways resistance and pulmonary vascular resistance seen in CLD. PAF is proinflammatory causing further recruitment and activation of inflammatory cells. At least two authors have found evidence of increased PAF in tracheal effluent from infants who develop CLD [11-13].

One of the mechanisms for closely regulating the expression of PAF is through the enzyme responsible for its degradation, PAF-acetylhydrolase (PAF-AH). PAF-AH is a phospholipase that is specific for PAF and PAF-like lipids. Acquired deficiencies in PAF-AH activity have been implicated in a variety of inflammatory conditions, including asthma. In addition to acquired deficiencies, Miwa et al described an inherited form of PAF-AH deficiency in the Japanese population [14]. Stafforini et al, at the University of Utah, cloned the PAF-AH gene and described a point mutation in the gene that explains this inherited PAF-AH deficiency [1, 2]. In studies of Japanese patients, they found that the PAF-AH gene was a modulating locus for severity of asthma. Recently, other variants of the PAF-AH gene have been found to be associated with inflammatory diseases, in particular asthma, in Caucasian populations [3].

A study performed in twins revealed a possible genetic susceptibility to chronic lung disease of prematurity [15]. It is possible that genetic alterations in pro and anti-inflammatory gene may contribute to a predisposition to the development of chronic lung disease. It is not known whether inherited deficiencies in PAF-AH activity may contribute to CLD. This study would begin to address the possibility of genetic factors that predispose to the development of CLD in preterm infants.

If the results of this observational study show an association between inherited or developmental deficiencies of PAF-AH activity and the development of CLD, a prospective randomized clinical trial of treatment with recombinant PAF-AH to prevent CLD might be considered.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in the NICU who:

  1. weigh ≤ 1500 grams at birth,
  2. are enrolled at age ≤ 5 days,
  3. require mechanical ventilation or continuous positive airway pressure (CPAP),
  4. have parents or guardians that have signed the informed consent document.

Exclusion Criteria:

* Infants with major congenital anomalies will be excluded.

Max Age: 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Eligible Patients
  Patients hospitalized in the NICU who:
  1. weigh ≤ 1500 grams at birth,
  2. are enrolled at age ≤ 5 days,
  3. require mechanical ventilation or continuous positive airway pressure (CPAP),
  4. have parents or guardians that have signed the informed consent document. Excluded Patients Infants with major congenital anomalies will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2002-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Chronic Lung Disease (CLD) and survival at 36 weeks corrected gestational age (CGA). | at 36 weeks (CGA)
  CLD will be defined as an oxygen requirement and abnormal x-ray findings. Investigations will compare outcomes of participants with genotypic variants of PAF-AH and those without known PAF-AH polymorphisms. Also, participant with biochemical evidence of PAF-AH dysregulation will be compared to those with normal PAF-AH protein and PAF concentrations.

SECONDARY OUTCOMES:
PAF-AH genotypic and phenotypic status in relation to multiple morbidities associated with prematurity. | 18 months
  The following clinical data will be collected and evaluated with respect to PAF-AH genotypic and phenotypic status: 1) length of time on mechanical ventilation; 2) length of time on oxygen therapy; 3) documented episodes of infection; 4) hemodynamically significant patent ductus arteriosus (PDA); 5) necrotizing enterocolitis (NEC); 6) retinopathy of prematurity (ROP); 7) intraventricular hemorrhage (IVH); 8) periventricular leukomalacia (PVL); 9) length of hospitalization; and 10) neurodevelopmental outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Christian C Yost, M.D., Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of Utah, Salt Lake City, Utah
  - Primary Children's Medical Center, Salt Lake City, Utah